CLINICAL TRIAL: NCT02731534
Title: Phase III Study of Z-213 in Subjects With Iron-deficiency Anemia
Brief Title: Efficacy Study of Intravenous Iron Preparation to Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z213-02
Record Dates: First submitted 2016-04-03; First posted 2016-04-07 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2017-01

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z-213 (Experimental)
  Interventions: Drug: Z-213
- Saccharated Ferric Oxide (Active Comparator)
  Interventions: Drug: Saccharated Ferric Oxide

INTERVENTIONS:
Drug: Z-213 — The total iron dosage is calculated based on hemoglobin value and the patients' weight, IV on day 1, 8 and 15 (if needed)
  Arms: Z-213
Drug: Saccharated Ferric Oxide — The total iron dosage is calculated based on hemoglobin value and the patients' weight, IV two or three times per week
  Arms: Saccharated Ferric Oxide

SUMMARY:
The purpose of this study is to confirm the non-inferiority of Z-213 compared to Saccharated Ferric Oxide using the maximum change in Hb from baseline over 12 weeks in patients with Iron-deficiency Anemia (IDA)

ELIGIBILITY:
Inclusion Criteria:

* Patients with iron deficiency anemia

Exclusion Criteria:

* Patients with anemia caused by conditions other than iron deficiency
* Patients with abnormal laboratory test values at screening for Serum phosphorus, Aspartate aminotransferase, Alanine aminotransferase
* Patients with liver, kidney or circulatory system disease
* Patients with a history or present illness that is a malignant tumor or autoimmune disease
* Patients who underwent intravenous administration of an iron preparation, administration of an erythropoiesis stimulation agent or blood transfusion within 8 weeks before the screening
* Patients who underwent oral administration of an iron preparation (including an over-the-counter drug or supplement) within 4 weeks before the screening

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Maximum change in Hb value | 12 weeks

SECONDARY OUTCOMES:
Change in Hb value | 12 weeks
Proportion of responders | 12 weeks
Proportion of subjects with normalization in Hb value | 12 weeks
Proportion of cumulative dosage | 12 weeks
Dosing period and the number of doses | 12 weeks
Incidence of Adverse Events | 12 weeks
Incidence of Adverse Drug Reactions | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan